CLINICAL TRIAL: NCT03168412
Title: A Study on Immunogenicity of Recombinant Hepatitis E Vaccine (Escherichia Coli) Hecolin® Using Accelerated Vaccination Schedule in Adults (Aged Over 18 Years)
Brief Title: A Study on the Recombinant Hepatitis E Vaccine (Escherichia Coli) (Accelerated Vaccination Schedule)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Xiamen Innovax Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRO-HE-008
Record Dates: First submitted 2017-05-14; First posted 2017-05-30 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Hepatitis E
Keywords: Hepatitis E
MeSH Terms: conditions — Hepatitis E | interventions — hecolin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the Accelerated Vaccination Schedule Group (Experimental): Participants in this arm are aged over 18 years and would receive three doses of Recombinant Hepatitis E Vaccine (Escherichia Coli)(Hecolin®) at 0,7,21 day.
  Interventions: Biological: Recombinant Hepatitis E Vaccine (Escherichia Coli)
- the Standard Vaccination Schedule Group (Active Comparator): Participants in this arm are aged over 18 years and would receive three doses of Recombinant Hepatitis E Vaccine (Escherichia Coli)(Hecolin®) at 0,1,6 month.
  Interventions: Biological: Recombinant Hepatitis E Vaccine (Escherichia Coli)

INTERVENTIONS:
Biological: Recombinant Hepatitis E Vaccine (Escherichia Coli) — Participants would receive 3 doses of Recombinant Hepatitis E Vaccine (Escherichia Coli) intramuscularly at 0, 7, 21 days.
  Other Names: Hecolin®
  Arms: the Accelerated Vaccination Schedule Group
Biological: Recombinant Hepatitis E Vaccine (Escherichia Coli) — Participants would receive 3 doses of Recombinant Hepatitis E Vaccine (Escherichia Coli) intramuscularly at 0, 1, 6 month.
  Other Names: Hecolin®
  Arms: the Standard Vaccination Schedule Group

SUMMARY:
This phase IV clinical study was designed to evaluate the immunogenicity and safety of the recombinant Hepatitis E vaccine (Hecolin®), manufactured by Xiamen Innovax Biotech CO., LTD., in healthy adults (over 18 years) with accelerated vaccination schedule. The study volunteers will receive the 3 doses of Hecolin® administered intramuscularly according to a 0-7-21 days schedule or a 0-1-6 month schedule.

ELIGIBILITY:
Inclusion Criteria:

1. Aged over 18 years old on the day of enrollment, including 18 years old;
2. Axillary temperature is below than 37.0 ℃;
3. Negative serological markers for hepatitis E and liver function are normal or no clinical significance;
4. Judged as healthy and eligible for vaccination by the investigators through a selfreported medical history and some physical examinations;
5. Able to understand this study information and willing to comply with all study requirements;
6. Willing to participate in this study and sign informed consent form.

Exclusion Criteria:

1. Pregnancy,breast-feeding or plan to be pregnant in 7 months;
2. Administration of Hepatitis E Vaccine before the study;
3. Participate in any other clinical trial during the study period;
4. Use of any investigational product or non-registered product (drug or vaccine)within 30 days preceding the first dose of the study vaccine or plan to use during the study period;
5. Received immunosuppressed, immunoregulation therapy or corticosteroid systemic therapy for more than 14 days in the 6 months before entry, except local treatment;
6. Administration of any immunoglobulin or blood products within 3 months preceding the first dose of the study vaccine,or plan to use during the study period;
7. Administration of any inactivated vaccines within 14 days preceding the first dose of the study or attenuated live vaccines within 21 days preceding the first dose of the study;
8. Had a fever (axillary temperature over 38°C) within 3 days or acute illness, or use systemic antibiotics or antiviral treatment within 5 days before vaccination;
9. Immunodeficiency (such as HIV carriers), primary disease of important organs, malignant tumor, or any immune disease (such as systemic lupus erythematosus, arthritis pauperum, splenectomy or functional asplenia or other disease which might affect immune response), liver and kidney disease and other chronic disease history;
10. History of allergic disease or history of serious adverse events occurring after vaccination, i.e., allergy,urticaria, dyspnea, angioneurotic edema or abdominal pain. Allergic history to any component of this vaccine.
11. Asthma that needed emergency treatment, hospitalization, oral or intravenous corticosteroid to keep stable in the past two years;
12. Combining another severe internal medicine disease(such as cardiopathy,diabetes and hyperthyroidism)
13. Anormal coagulation function or coagulopathy diagnosed by doctor;
14. Epilepsy(not including alcohol epilepsy within 3 years prior to abstinence and simple epilepsy that do without curing within 3 years prior to the study )
15. Anomal psychology or mind affecting the individual's ability to obey the study requirement;
16. Other medical, psychological, social or occupational factors that, according to the investigators' judgment,might affect the individual's ability to obey the protocol or sign the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2017-05-25 (Actual); Primary Completion 2018-07-15 (Actual); Study Completion 2018-11-28 (Actual)

PRIMARY OUTCOMES:
Anti-HEV antibody of Experimental Group | up to 2 months
  Measure anti-HEV antibody in serum samples at 51st day to evaluate the immunogenicity of the Hepatitis E vaccine.

SECONDARY OUTCOMES:
Adverse reactions/events of Experimental Group and Control Group | up to 7 months
  Measure solicited local adverse reactions/events within 7 days after each vaccination; Measure solicited systematic adverse reactions/events within 7 days after each vaccination; Measure unsolicited adverse reactions/events within 30 days after vaccination; Measure serious adverse events occurred throughout the study（up to 7 months）.
Anti-HEV antibody of Experimental Group | up to 7 months
  Measure anti-HEV antibody in serum samples at 21st day,28st day and month 7 to evaluate the immunogenicity of the Hepatitis E vaccine.
Anti-HEV antibody of Control Group | up to 7 months
  Measure anti-HEV antibody in serum samples at month 1,2,7 to evaluate the immunogenicity of the Hepatitis E vaccine.

CONTACTS AND LOCATIONS:
Overall Officials: Zhiping Chen, Principal Investigator — Zhejiang Provincial Center for Disease Control and Prevention
Locations (1):
- Changshan Center for Disease Control and Prevention, Quzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen Z, Lin S, Duan J, Luo Y, Wang S, Gan Z, Yi H, Wu T, Huang S, Zhang Q, Lv H. Immunogenicity and safety of an accelerated hepatitis E vaccination schedule in healthy adults: a randomized, controlled, open-label, phase IV trial. Clin Microbiol Infect. 2019 Sep;25(9):1133-1139. doi: 10.1016/j.cmi.2019.01.015. Epub 2019 Jan 31. PMID 30711651